CLINICAL TRIAL: NCT07218432
Title: A Window of Opportunity Pilot Study: TheraBionic P1 Device for Patients With Resectable Early-stage Breast Cancer in a Neoadjuvant Setting
Brief Title: A Study of the TheraBionic P1 Device in Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Lubina Arjyal MD, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-026
Record Dates: First submitted 2025-09-09; First posted 2025-10-20 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer Stage I; Breast Cancer Stage II; Breast Cancer Stage IIIA; Hormone Receptor Positive Tumor; HER2-negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- TheraBionic P1 device (Experimental): Self Administered Amplitude-modulated electromagnetic fields three times daily
  Interventions: Device: TheraBionic P1 Device

INTERVENTIONS:
Device: TheraBionic P1 Device — Amplitude-modulated electromagnetic fields will be self-administered and given continuously to patients in three 60-minute treatments per day, administered in the morning, middle of the day and in the evening prior to surgical resection of early stage breast cancer.

SUMMARY:
The goal of this clinical trial is to learn if adding cancer-specific amplitude-modulated radiofrequency electromagnetic field therapy (TheraBionic P1 device) to the treatment of resectable early-stage breast cancer will affect the pathological response.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have histologically proven invasive breast cancer that is HR (hormone receptor) positive and HER2 (Human Epidermal Growth Factor Receptor 2) negative according to the 2010 American Society of Clinical Oncology (ASCO) College of American Pathologists (CAP) guidelines (ER and/or PR (progesterone receptor) >1% and HER2 negative by immunohistochemistry [IHC] and/or fluorescent in situ hybridization [FISH]).
* Participant must have early-stage operable disease (stage I-II or III who have planned upfront surgery) and agree to definitive upfront surgery.
* Participant must be available for at least two weeks of TheraBionic treatment prior to scheduled resection
* Participant must have archival tissue available.
* Participant must be a woman aged 22 years or older
* Participant must be able to understand a written informed consent document and be willing to sign it
* Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* It is not known what effects this treatment has on human pregnancy or development of the embryo or fetus. Therefore, women of child-bearing potential must agree to avoid becoming pregnant starting at initiation of treatment up until at least 30 days after the last TheraBionic P1 session

Exclusion Criteria:

* Participants that are receiving or will receive neoadjuvant chemotherapy or neoadjuvant hormonal therapy
* Participants with known active secondary malignancy, unless, in the opinion of the investigator, it is unlikely to interfere with the safety and efficacy of the endpoints
* Participants that are taking any other investigational drugs
* Participants that are pregnant or breastfeeding due to the unknown but potential risk for adverse events. If a breastfeeding participant would like to be part of this study, breastfeeding must be discontinued
* Participants with active oral mucosal inflammation, ulceration, or other pathology that could interfere with the use of TheraBionic P1 device (for example: mucositis, thrush, bleeding mucosal lesions, oral herpes, aphthous stomatitis, mouth ulcers, chancre sores, gingivostomatitis, herpangina, aphthae).
* Participants receiving calcium channel blockers and any agent blocking L-type or T-type voltage gated calcium channels (for example: amlodipine, nifedipine, ethosuximide, ascorbic acid/vitamin C, etc.) unless their medical treatment is discontinued at least one day prior to treatment. Participant must agree to abstain from using calcium channel blockers for the duration of treatment on study.
* Participants that do not agree to be followed according to the study protocol or have cognitive or physical inability to use the device

Min Age: 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-10 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Pathological Response to Treatment | At time of surgery (after approximately 2 weeks of treatment and tumor resection)
  Proportion of responders based on residual cancer cells in a resection specimen will be quantified. The response rate will be estimated as the proportion of patients who respond to treatment relative to all patients. The corresponding two-sided 95% confidence interval (CI) will be calculated using Clopper and Pearson's method

SECONDARY OUTCOMES:
Changes in microRNA expression in tumor tissue | Baseline to post-surgical resection
  Changes in microRNA expression in tumor tissue pre- and post-treatment will be calculated as the difference between pre- and post-treatment expression values with two-sided 95% CI estimated using a standard t-distribution-based formula for paired differences.
Changes in Ki-67 expression in tumor tissue | Baseline to post-surgical resection
  Changes in Ki-67 expression in tumor tissue pre- and post-treatment will be calculated as the difference between pre- and post-treatment expression values with two-sided 95% CI estimated using a standard t-distribution-based formula for paired differences.
Changes in tumor apoptosis marker Cleaved caspase-3 (CC3) in tumor tissue | Baseline to post-surgical resection
  Changes in CC3 expression in tumor tissue pre- and post-treatment will be calculated as the difference between pre- and post-treatment expression values with two-sided 95% CI estimated using a standard t-distribution-based formula for paired differences.
Changes in cell cycle arrest marker p27 in tumor tissue | Baseline to post-surgical resection
  Changes in p27 expression in tumor tissue pre- and post-treatment will be calculated as the difference between pre- and post-treatment expression values with two-sided 95% CI estimated using a standard t-distribution-based formula for paired differences.
Overall survival (OS) | Up to 5 years post-surgery
  OS will be graphically summarized using Kaplan-Meier (KM) curves, with corresponding medians and two-sided 95% CIs computed using KM estimates. Additionally, OS rates at every six months post-treatment will be estimated using the KM estimated, with two-sided 95% CIs provided for each time point.
Progression Free Survival (PFS) | Up to 5 years post-surgery
  PFS will be graphically summarized using Kaplan-Meier (KM) curves, with corresponding medians and two-sided 95% CIs computed using KM estimates. Additionally, PFS rates at every six months post-treatment will be estimated using the KM estimated, with two-sided 95% CIs provided for each time point.

OTHER OUTCOMES:
Positron Emission Tomography with 3'-Deoxy-3'-18F-Fluorothymidine (PET-FLT) association of response to treatment | From Screening to after 7 days of treatment with the TheraBionic Device.
  Changes in the SUV max as measured by FLT-PET prior to treatment compared to after treatment and before resection. SUV (standard uptake value) max values will be log-transformed and descriptively summarized using the mean, standard deviation, and two-sided 95% CI. Changes in SUV max pre- and post-treatment will be calculated as the difference between the pre- and post-treatment values with two-sided 95% CI estimated using a standard t-distribution-based formula for paired differences. The association between changes in SUV max and response will be explored using logistic regression analysis. Optional study for the first 5 participants.

CONTACTS AND LOCATIONS:
Overall Officials: Lubina Arjyal, M.D., Principal Investigator — Wayne State University
Locations (1):
- Karmanos Cancer Institute, Detroit, Michigan, United States